CLINICAL TRIAL: NCT00204711
Title: Use of the SNAP II EEG Monitor in Outpatients Undergoing Surgery/Procedures With Sedation
Brief Title: Use of the SNAP II Electroencephalography (EEG) Monitor in Outpatients Undergoing Surgery/Procedures With Sedation
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2005-0014; SNAPII
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Sedation
Keywords: patients having outpatient surgery with sedation; patients having procedures with sedation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outpatient Surgery with Sedation: SNAP II EEG data will be recorded continuously during the sedation and intermittently compared to routinely monitored parameters of sedation adequacy including vital signs, patient movement, grimacing, verbal complaints, and patient responsiveness to verbal and tactile stimuli. Following surgery, patients will be questioned to determine recall or memory of discomfort.
  Interventions: Other: SNAP II EEG System

INTERVENTIONS:
Other: SNAP II EEG System — A portable EEG monitor (SNAP II EEG System, Everest -St. Louis) is unique in that it monitors both low frequency EEG signals (1-40 Hz), which are typically used, and high frequency EEG signals (80-420 Hz), which are not usually used, and calculates a derived EEG parameter (the SNAP Index). The SNAP Index ranges from 100 (completely awake) to 0 (no brain activity) and has been shown in a few studies to correlate with increasing sedation and loss of consciousness in human volunteers and patients receiving general anesthesia during surgery.

SUMMARY:
The purpose of this study is to determine if the SNAP II electroencephalography (EEG) monitor accurately reflects changes in sedation level in outpatients undergoing surgery or procedures with sedation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I, II or III physical status

Exclusion Criteria:

* Use of inhalation general anesthesia
* ASA IV physical status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing outpatient (same day) surgery/procedures with sedation
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2005-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Assessment of participant heterogeneity between SNAP Index and OASS Score. | up to 1 day post op
  The SNAP Index is a derived EEG (electroencephalogram) parameter (from the SNAP II EEG System) ranging from 100 (completely awake) to 0 (no brain activity). The Observer's Assessment of Alertness/Sedation Score (OASS) is a score derived from motor and sensory functions between 0 and 5 where 0 is unresponsive and 5 is awake.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Springman, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Springman SR, Andrei AC, Willmann K, Rusy DA, Warren ME, Han S, Lee M. A comparison of SNAP II and bispectral index monitoring in patients undergoing sedation. Anaesthesia. 2010 Aug;65(8):815-9. doi: 10.1111/j.1365-2044.2010.06408.x. Epub 2010 Jun 25. PMID 20586747